CLINICAL TRIAL: NCT05436418
Title: Phase I/II Trial to Determine the Lowest Effective Dose of Post-Transplantation Cyclophosphamide in Combination With Sirolimus and Mycophenolate Mofetil as Graft-Versus-Host Disease Prophylaxis After Reduced Intensity Conditioning and Peripheral Blood Stem Cell Transplantation
Brief Title: The Lowest Effective Dose of Post-Transplantation Cyclophosphamide in Combination With Sirolimus and Mycophenolate Mofetil as Graft-Versus-Host Disease Prophylaxis After Reduced Intensity Conditioning and Peripheral Blood Stem Cell Transplantation
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 10000613; 000613-C
Record Dates: First submitted 2022-06-24; First posted 2022-06-29 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12-11

CONDITIONS: Peripheral Blood Stem Cell Transplantation; Hematopoietic Stem Cell Transplantation
Keywords: Reduced Intensity Conditioning; Systemic Immunosuppressive Therapy; Hematologic Malignancy; Acute Myeloid Leukemia; Calcineurin Inhibitor
MeSH Terms: conditions — Hematologic Neoplasms; Leukemia, Myeloid, Acute | interventions — Melphalan; Sirolimus; Whole-Body Irradiation; Cyclophosphamide; fludarabine; Mesna; Filgrastim

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Donors (Haplo HCT) (No Intervention): Research on collected samples
- Donors (Matched HCT) (No Intervention): Research on collected samples
- Phase I Dose De-escalation (Haplo HCT) (Experimental): PTCy at de-escalating doses to assess for safety and determine Phase II dose
  Interventions: Drug: Melphalan; Drug: Sirolimus; Radiation: Total Body Irradiation (TBI); Drug: Cyclophosphamide; Drug: Mycophenolate Mofeti; Drug: Fludarabine; Procedure: Allogeneic HSCT; Drug: Mesna; Drug: Filgrastim
- Phase I Dose De-escalation (Matched HCT) (Experimental): PTCy at de-escalating doses to assess for safety and determine Phase II dose
  Interventions: Drug: Melphalan; Drug: Sirolimus; Radiation: Total Body Irradiation (TBI); Drug: Cyclophosphamide; Drug: Mycophenolate Mofeti; Drug: Fludarabine; Procedure: Allogeneic HSCT; Drug: Mesna; Drug: Filgrastim
- Phase I Pilot for Comparative Data (Haplo HCT) (Experimental): Standard PTCy 50 mg/kgday on days +3 and +4
  Interventions: Drug: Melphalan; Drug: Sirolimus; Radiation: Total Body Irradiation (TBI); Drug: Cyclophosphamide; Drug: Mycophenolate Mofeti; Drug: Fludarabine; Procedure: Allogeneic HSCT; Drug: Mesna; Drug: Filgrastim
- Phase I Pilot for Comparative Data (Matched HCT) (Experimental): Standard PTCy 50 mg/kg/day on days +3 and +4
  Interventions: Drug: Melphalan; Drug: Sirolimus; Radiation: Total Body Irradiation (TBI); Drug: Cyclophosphamide; Drug: Mycophenolate Mofeti; Drug: Fludarabine; Procedure: Allogeneic HSCT; Drug: Mesna; Drug: Filgrastim
- Phase II Efficacy (Haplo HCT) (Experimental): PTCy at shortest duration, safe dose (from Phase I)
  Interventions: Drug: Melphalan; Drug: Sirolimus; Radiation: Total Body Irradiation (TBI); Drug: Cyclophosphamide; Drug: Mycophenolate Mofeti; Drug: Fludarabine; Procedure: Allogeneic HSCT; Drug: Mesna; Drug: Filgrastim
- Phase II Efficacy (Matched HCT) (Experimental): PTCy at shortest duration, safe dose (from Phase I)
  Interventions: Drug: Melphalan; Drug: Sirolimus; Radiation: Total Body Irradiation (TBI); Drug: Cyclophosphamide; Drug: Mycophenolate Mofeti; Drug: Fludarabine; Procedure: Allogeneic HSCT; Drug: Mesna; Drug: Filgrastim

INTERVENTIONS:
Drug: Melphalan — Matched HCT: 100 mg/m^2 IV on day -2 over 30 minutes. Haplo HCT:
  100 mg/m^2 IV on day -6 over approximately 20-30 minutes.
  Arms: Phase I Dose De-escalation (Haplo HCT); Phase I Dose De-escalation (Matched HCT); Phase I Pilot for Comparative Data (Haplo HCT); Phase I Pilot for Comparative Data (Matched HCT); Phase II Efficacy (Haplo HCT); Phase II Efficacy (Matched HCT)
Drug: Sirolimus — Sirolimus: Loading dose of 6 mg orally given on day +5 (calculated based on actual body weight, max initial dose 6 mg)^d, then maintenance dose starting at 2 mg orally daily on day +6 with dose adjustments to maintain a trough of 5-12 ng/ml, continued through day +80 with no taper. Doses should be modified as appropriate for drug interactions and may be modified based on institutional practice.
  Arms: Phase I Dose De-escalation (Haplo HCT); Phase I Dose De-escalation (Matched HCT); Phase I Pilot for Comparative Data (Haplo HCT); Phase I Pilot for Comparative Data (Matched HCT); Phase II Efficacy (Haplo HCT); Phase II Efficacy (Matched HCT)
Radiation: Total Body Irradiation (TBI) — Haplo HCT only: A dose of 200 cGy will be administered on day -1.
  Arms: Phase I Dose De-escalation (Haplo HCT); Phase I Dose De-escalation (Matched HCT); Phase I Pilot for Comparative Data (Haplo HCT); Phase I Pilot for Comparative Data (Matched HCT); Phase II Efficacy (Haplo HCT); Phase II Efficacy (Matched HCT)
Drug: Cyclophosphamide — based on dose level being tested (50, 35, 25, or 15 mg/kg) IV once daily over 2 hours on days +3 and +4. Cyclophosphamide will be dosed according to ideal body weight. Cyclophosphamide infusion on days +3 should be started between 70-74 hours after the start of the PBSC infusion. Cyclophosphamide infusion on day +4 should be started between 94-98 hours after the start of the bone marrow infusion.
  Arms: Phase I Dose De-escalation (Haplo HCT); Phase I Dose De-escalation (Matched HCT); Phase I Pilot for Comparative Data (Haplo HCT); Phase I Pilot for Comparative Data (Matched HCT); Phase II Efficacy (Haplo HCT); Phase II Efficacy (Matched HCT)
Drug: Mycophenolate Mofeti — 15 mg/kg orally or IV three times daily (max 1000 mg/dose) starting on day +5, continued through day +35. Dosing will be according to actual body weight.
  Arms: Phase I Dose De-escalation (Haplo HCT); Phase I Dose De-escalation (Matched HCT); Phase I Pilot for Comparative Data (Haplo HCT); Phase I Pilot for Comparative Data (Matched HCT); Phase II Efficacy (Haplo HCT); Phase II Efficacy (Matched HCT)
Drug: Fludarabine — Matched HCT: 25 mg/m^2/day infused IV over 60 minutes from day -7 to day -3. Haplo HCT: 40 mg/m^2/day infused IV over approximately 30-60 minutes from day -5 to day -2
  Arms: Phase I Dose De-escalation (Haplo HCT); Phase I Dose De-escalation (Matched HCT); Phase I Pilot for Comparative Data (Haplo HCT); Phase I Pilot for Comparative Data (Matched HCT); Phase II Efficacy (Haplo HCT); Phase II Efficacy (Matched HCT)
Procedure: Allogeneic HSCT — Stem cell transplant
  Arms: Phase I Dose De-escalation (Haplo HCT); Phase I Dose De-escalation (Matched HCT); Phase I Pilot for Comparative Data (Haplo HCT); Phase I Pilot for Comparative Data (Matched HCT); Phase II Efficacy (Haplo HCT); Phase II Efficacy (Matched HCT)
Drug: Mesna — equal to the cyclophosphamide dose (50, 35, 25, or 15 mg/kg) as IV infusion concomitant with cyclophosphamide. Mesna is dosed in the same way as cyclophosphamide regarding ideal vs. actual body weight.b Dosing may be modified based on institutional standard practice.
  Arms: Phase I Dose De-escalation (Haplo HCT); Phase I Dose De-escalation (Matched HCT); Phase I Pilot for Comparative Data (Haplo HCT); Phase I Pilot for Comparative Data (Matched HCT); Phase II Efficacy (Haplo HCT); Phase II Efficacy (Matched HCT)
Drug: Filgrastim — begins on day +5 at a dose of 5 mcg/kg/day (actual body weight; dose rounding is permitted e.g., nearest vial or syringe size) and is administered daily subcutaneously or IV until the absolute neutrophil count is > 1000 cells/mm3 for three days or > 5000 for one day.
  Arms: Phase I Dose De-escalation (Haplo HCT); Phase I Dose De-escalation (Matched HCT); Phase I Pilot for Comparative Data (Haplo HCT); Phase I Pilot for Comparative Data (Matched HCT); Phase II Efficacy (Haplo HCT); Phase II Efficacy (Matched HCT)

SUMMARY:
Background:

Blood cancers (such as leukemias or lymphomas) often do not respond to standard treatments. A transplant of blood stem cells from a healthy donor can help people with these cancers. Sometimes these transplants cause serious side effects, including a common immunologic problem called graft-versus-host disease. A drug called cyclophosphamide given early after the transplant (post-transplantation cyclophosphamide, PTCy) can reduce these complications. But sometimes this drug has its own negative effects. Furthermore, studies in mice suggest that an intermediate, rather than very high, dose of this drug may best protect against graft-versus-host disease.

Objective:

To find out if a lower dose of PTCy is more helpful for people who undergo blood stem cell transplants.

Eligibility:

People aged 18 and older who have a blood cancer and are eligible for a transplant of blood stem cells from another person. Healthy donors are also needed but must be related to the individual needing the transplant.

Design:

Participants will undergo screening. Transplant recipients will have imaging scans and tests of their heart and lung function. They will be assessed for the status of their cancer, including bone marrow taken from their pelvis and possibly also scans and/or fluid drawn from the spine depending on the disease type.

Donors will be screened for general health. They will give several tubes of blood. They will give an oral swab and saliva and stool samples for research.

Recipients will be in the hospital at least 4 to 6 weeks.

They will have a temporary catheter inserted into a vein in the chest or neck. Medications will be given and blood will be drawn through the catheter.

The transplanted stem cells will be given through the catheter. Participants will receive medications both before and after the transplant.

Participants will return to the clinic at least once a week for 3 months after leaving the hospital. Follow-up visits will continue periodically for 5 years.

DETAILED DESCRIPTION:
Background:

* Post-transplantation cyclophosphamide (PTCy) reduces rates of severe acute and chronic graft-versus-host disease (GVHD) after allogeneic hematopoietic cell transplantation (HCT) and safely facilitates human leukocyte antigen (HLA)-haploidentical HCT
* When clinically translated, the dose (50 mg/kg) and timing (days +3 and +4) of PTCy used were partly extrapolated from murine major histocompatibility complex (MHC)-matched skin allografting models and were partly empirical
* In both MHC-haploidentical and MHC-disparate murine HCT models, a dose of 25 mg/kg/day was superior to 50 mg/kg/day on days +3 and +4 in terms of protection against GVHD severity and mortality. Lower dosing of PTCy also was associated with less broad reduction of T-cell numbers after PTCy and lower toxicity than higher dosing.
* In patients on an NIH study using myeloablative conditioning and bone marrow as the graft source, a dose of 25 mg/kg/day on days +3/+4 has been associated with more rapid engraftment, less toxicity, and potentially better immune function without an increase in acute GVHD.
* The optimal dosing of PTCy potentially may differ depending on the graft source (bone marrow versus peripheral blood stem cells) and HLA disparity (HLA-matched vs. HLA-partially mismatched).

Objective:

* Phase I: Determine the lowest effective dose of post-transplantation cyclophosphamide (PTCy) in combination with sirolimus and mycophenolate mofetil (MMF) as graft-versus-host disease (GVHD) prophylaxis after reduced intensity conditioning and peripheral blood stem cell transplantation (PBSCT), as assessed by primary graft failure AND Grade III-IV acute GVHD as the dose limiting toxicities (DLTs). This lowest effective dose will be evaluated in parallel for HLA-matched and HLA-haploidentical HCT in different arms of the study.
* Phase II: Evaluate the efficacy of PTCy, at the lowest dose determined for each HLA-matching arm from phase I, as assessed by 1-year GVHD-free relapse-free survival (GRFS) rate.

Eligibility:

-Recipient Participant:

* Histologically or cytologically confirmed hematologic malignancy with standard indication for allogeneic hematopoietic cell transplantation
* Age >= 50 years or 18-49 years but considered ineligible for myeloablative conditioning.
* At least one potentially suitable HLA-haploidentical or 10/10 (HLA-A, B, C, DR, DQ) related or unrelated donor.
* Karnofsky performance score >= 70
* Adequate organ function

Design:

* Open-label, multi-center, non-randomized, phase I/II study.
* All recipient participants will receive reduced intensity conditioning, peripheral blood stem cell (PBSC) HCT, and GVHD prophylaxis with PTCy, MMF, and sirolimus.
* There will be two parallel arms: one using HLA-haploidentical donors and one using HLA-matched related or unrelated donors.
* A small pilot of 10 evaluable participants per arm will receive the standard PTCy 50 mg/kg/day on days +3/+4 to obtain a limited amount of comparative clinical, pharmacokinetic, and T-cell immunophenotyping data.
* The study will proceed to a novel phase I time-to-event Bayesian optimal interval (TITE-BOIN) trial design to find the lowest acceptable dose of PTCy for each arm. Primary graft failure and grade III-IV aGVHD at day +100 post-transplant are defined PTCy dose-limiting toxicities.
* Three dose levels of PTCy: 35, 25, and 15 mg/kg/day on days +3 and +4 are planned in each arm of phase I.
* Recipient participants will be evaluated for development of grade III-IV acute GVHD (aGVHD) and primary graft failure at day +100 as the dose-limiting toxicities. Once the optimal PTCy dose for PBSC transplantation is determined for each arm, we will conduct a phase II expansion for each arm to estimate the efficacy of PTCy in combination with sirolimus and mycophenolate mofetil as GVHD prophylaxis. 1-year GRFS rate will be the primary endpoint during the phase II part.

ELIGIBILITY:
* INCLUSION CRITERIA:

Recipient

* Participants must have a histologically or cytologically confirmed hematologic malignancy with standard indication for allogeneic hematopoietic cell transplantation limited to one of the following:

  * Acute myeloid leukemia (AML) of intermediate or adverse risk disease by the 2017 European LeukemiaNet criteria in first morphologic complete remission (<5% blasts in the bone marrow, no detectable abnormal peripheral blasts, and no extramedullary disease)
  * AML of any risk in second or subsequent morphologic complete remission
  * Acute lymphoblastic leukemia in first or subsequent complete remission
  * Myelodysplastic syndrome of intermediate or higher score by the Revised International Prognostic Scoring System (IPSS-R)
  * Primary myelofibrosis of intermediate-2 or higher risk by the DIPSS
  * Chronic myelomonocytic leukemia
  * Chronic myelogenous leukemia resistant to or intolerant of >= 3 tyrosine kinase inhibitors or with history of accelerated phase or blast crisis
  * B-cell lymphoma including Hodgkin lymphoma that has relapsed within 1 year of completion of primary treatment, relapsed after autologous transplantation, or has progressed through at least 2 lines of therapy
  * Chronic lymphocytic leukemia with 17p deletion and/or unmutated IgHV or refractory to or intolerant of both BTK and PI3K inhibitors
  * Mature T or NK neoplasms as defined in the WHO guidelines of sufficient type and severity for allogeneic HCT based on the Prognostic Index for T-cell lymphoma (PIT) score of low-intermediate risk or higher or on recently published clinical practice guidelines
  * Hematologic malignancy of dendritic cell or histiocytic cell type
  * Multiple myeloma, stage III, relapsing after therapy with both a proteasome inhibitor and an immunomodulatory drug (IMiD)
* Age >= 50 years or age 18-49 years and also meeting one of the following criteria:

  * Prior myeloablative HCT
  * Prior exposure to inotuzumab, gemtuzumab, or other agent that increases the risk for sinusoidal obstruction syndrome.
  * Hematopoietic Cell Transplantation- Comorbidity Index (HCT-CI) >= 3
  * Karnofsky performance score <80
  * Co-morbidity considered by the treating physician to be exclusionary of myeloablative conditioning
* At least one potentially suitable HLA-haploidentical or 10/10 (HLA-A, B, C, DR, DQ) related or unrelated donor for HCT
* Karnofsky performance score >= 70
* Adequate organ function defined as possessing all of the following:

  * Cardiac ejection fraction >= 45% by 2D ECHO;
  * Forced expiratory volume-1 (FEV-1), forced vital capacity (FVC), and diffusing capacity of the lung for carbon monoxide (DLCO) (corrected for hemoglobin) all of >= 50% predicted;
  * Estimated serum creatinine clearance of >= 60 ml/minute/1.73m^2 calculated using eGFR in the clinical lab;
  * Total bilirubin <= 2X the upper limit of normal;
  * Alanine aminotransferase and aspartate aminotransferase <= 3X the upper limit of normal.
* Individuals of child-bearing potential (IOCBP) and participants who can father children must agree to use highly effective contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for at least one year post-transplant.
* IOCBP must have a negative serum or urine pregnancy test within 7 days prior to initiation of conditioning regimen.
* Ability of participant to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

Recipient

* Participants who are receiving any other investigational agents. Prior experimental therapies must have been completed at least 2 weeks prior to the date of beginning conditioning.
* Active nursing.
* Active malignancy of non-hematopoietic type (excluding non-melanoma skin cancers) which is: metastatic, or relapsed/refractory to treatment, or locally advanced and not amenable to curative treatment, or limited disease treated with curative intent treatment within the last 2 years. This excludes non-melanoma skin cancers.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to study agents.
* Uncontrolled intercurrent illness (e.g., severe endocrinopathy, disseminated intravascular coagulation, profound electrolyte disturbance, active infectious hepatitis, uncontrolled dental infection) that in the opinion of the Site PI would make it unsafe to proceed with transplantation.

INCLUSION CRITERIA:

Donor

* Related (age >=12) and unrelated (age >=18) donors deemed eligible (i.e., evaluated at NIH, COH, and FHCC in accordance with existing institutional Standard Policies and Procedures or evaluated per the standards required by the IRB of the National Marrow Donor Program or applicable registry), and willing to donate research samples will be included.
* Ability of participant or parent/legal guardian to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

Donor

None

Ages: 12 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2022-11-18 (Actual); Primary Completion 2027-06-25 (Estimated); Study Completion 2028-06-25 (Estimated)

PRIMARY OUTCOMES:
Phase II: Evaluate the efficacy of PTCy, at the lowest dose determined for each HLA-matching arm from phase I, as assessed by 1-year GVHD-free relapse-free survival (GRFS) rate. | 1 year
  1-year GRFS and 95% CI per arm will be estimated using Kaplan-Meier curves.
Phase I: Determine the lowest effective dose of PTCy in combination with sirolimus and mycophenolate mofetil as GVHD prophylaxis after reduced intensity conditioning and PBSCT, as assessed by primary graft failure AND Grade III-IV acute GVHD as ... | 60 days
  Number of evaluable subjects and DLT will be summarized per dose level in each arm.

SECONDARY OUTCOMES:
Estimate rates of symptomatic BK virus cystitis. (Phase I and II) | 100 days
  To evaluate symptomatic BK virus cystitis using Kaplan-Meier curves or competing risk-based cumulative incidence curves as appropriate. For phase I, these analyses will be presented descriptively or as proportions of subjects experiencing the outcome.
Estimate rates of hematopoietic recovery/engraftment. (Phase I and II) | day 28, 42, and 100
  Rate and timing of neutrophil and platelet engraftment also will be evaluated descriptively, including fractions who attain each condition at day 28, 42, and 100, along with 95% confidence intervals. Ranges and medians will be calculated only in engrafting subjects.
Estimate rates of Grade II-IV and III-IV acute GVHD at 100 days (Phase I and II) | 100 days
  To evaluate for grades II-IV and III-IV acute GVHD at 100 days using Kaplan-Meier curves or competing risk-based cumulative incidence curves. Competing risks will include relapse/progression and NRM. For phase I, these analyses will be presented descriptively or as proportions of subjects experiencing an outcome.
Estimate non-relapse mortality at one year (Phase II only) | 1 year
  To evaluate non-relapse mortality at one year, estimates will be determined using competing risk-based cumulative incidence curves. Relapse and non-relapse mortality will be competing risks for each other.
Estimate overall survival and progression-free survival at one year (Phase II only) | 1 year
  To evaluate survival at one year, estimates will be determined using Kaplan-Meier curves.
Estimate incidence progression/relapse at one year (Phase II only) | 1 year
  To evaluate relapse at one year, estimates will be determined using Kaplan-Meier curves or competing risk-based cumulative incidence curves as appropriate. Relapse and non-relapse mortality will be competing risks for each other.
Describe and characterize cytokine release syndrome (CRS) (Phase I and II) | 1 year
  To evaluate CRS incidence, frequency and severity using Kaplan-Meier curves or competing risk-based cumulative incidence curves as appropriate. Relapse/progression and NRM will be competing risks.
Estimate rates of CMV reactivation requiring preemptive therapy. (Phase I and II) | 100 days
  To evaluate CMV reactivation requiring preemptive therapy using Kaplan-Meier curves or competing risk-based cumulative incidence curves as appropriate. Competing risks will include relapse/progression and NRM. For phase I, these analyses will be presented descriptively or as proportions of subjects experiencing an outcome.
Estimate rates of any chronic GVHD and moderate/severe chronic GVHD at one year (Phase I and II) | 1 year
  To evaluate for all chronic and moderate/severe chronic GVHD at one year using Kaplan-Meier curves or competing risk-based cumulative incidence curves. Competing risks will include relapse/progression and NRM. For phase I, these analyses will be presented descriptively or as proportions of subjects experiencing an outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher G Kanakry, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (2):
- United States (2):
  - City of Hope, Duarte, California
  - National Institutes of Health Clinical Center, Bethesda, Maryland

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request. @@@@@@@@@@@@In addition, all large scale genomic sequencing data will be shared with subscribers to dbGaP.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.@@@@@@@@@@@@Genomic data are available once genomic data are uploaded per protocol GDS plan for as long as database is active.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI.@@@@@@@@@@@@Genomic data are made available via dbGaP through requests to the data custodians.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_000613-C.html